CLINICAL TRIAL: NCT02259127
Title: A Randomised Trial of Dolutegravir (DTG)-Based Antiretroviral Therapy vs. Standard of Care (SOC) in Children With HIV Infection Starting First-line or Switching to Second-line ART
Brief Title: ODYSSEY (PENTA 20)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Program for HIV Prevention and Treatment (PHPT) (Unknown); ViiV Healthcare (Industry); MRC CTU at UCL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ODYSSEY (PENTA 20); 2014-002632-14 (EudraCT Number)
Record Dates: First submitted 2014-09-30; First posted 2014-10-08 (Estimated); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOC arm (Active Comparator): Standard of Care (SOC) for ODYSSEY A is defined as a PI or non nucleoside transcriptase inhibitors + 2 or 3 nucleoside transcriptase inhibitor SOC for ODYSSEY B is defined as a PI or non nucleoside transcriptase inhibitor+ 2 nucleoside transcriptase inhibitors
  Interventions: Drug: Standard of Care
- DTG arm (Experimental): DTG + 2 nucleoside transcriptase inhibitors
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir
  Other Names: DTG
  Arms: DTG arm
Drug: Standard of Care — PI or non nucleoside transcriptase inhibitors
  Other Names: SOC
  Arms: SOC arm

SUMMARY:
A new anti-HIV medicine (Dolutegravir) combined with 2 currently used anti-HIV medicines is non-inferior to the standard combination of medicines used in terms of efficacy and better in terms of toxicity.

DETAILED DESCRIPTION:
The ODYSSEY study was an international randomised trial evaluating dolutegravir based antiretroviral therapy (ART) versus standard of care in HIV-infected children aged less than 18 years who were starting first line treatment (ODYSSEY A) or switching to second line treatment (ODYSSEY B). Participants had visits 4 weeks and 12 weeks after randomisation and every 12 weeks subsequent of that. They were followed up for a minimum of 96 weeks. The primary objective of the study was to assess the difference in virological or clinical failure by 96 weeks between children receiving a DTG-based regimen and those on standard of care.

At the end of study visit for the randomised phase, children and carers were invited to consent to extended follow-up. Children's visit schedules and care were as per local clinic guidelines. Participants were followed up until July 2023 in this phase of the trial. The objectives of the extended follow-up were two-fold: 1. to provide safety data for ViiV Healthcare for participants who, in the opinion of the treating physician, continue to derive benefit from dolutegravir and receive dolutegravir from ViiV Healthcare where it was not available through their country's national HIV treatment programme; 2. to monitor long-term safety and effectiveness of dolutegravir versus standard of care.

ELIGIBILITY:
Inclusion Criteria:

ALL PATIENTS:

* Children ≥28 days and <18 years weighing ≥3kg with confirmed HIV-1 infection
* Parents/carers and children, where applicable, give informed written consent
* Girls aged 12 years or older who have reached menses must have a negative pregnancy test at screening and be willing to adhere to effective methods of contraception if sexually active
* Children with co-infections who need to start ART can be enrolled into ODYSSEY according to local/national guidelines
* Parents/carers and children, where applicable, willing to adhere to a minimum of 96 weeks' follow-up

  * Children weighing 3 to <14kg must be eligible and willing to participate in the Weight band (WB)-Pharmacokinetics (PK)1 substudy unless direct enrolment for the child's weight band has opened following the WB-PK1 substudy and/or dosing information has become available from the IMPAACT P1093 DTG dose-finding study.

ADDITIONAL CRITERIA FOR ODYSSEY A:

• Planning to start first-line ART

ADDITIONAL CRITERIA FOR ODYSSEY B:

* Planning to start second-line ART defined as either: (i) switch of at least 2 ART drugs due to treatment failure; or (ii) switch of only the third agent due to treatment failure where drug sensitivity tests show no mutations conferring Nucleoside Reverse Transcriptase Inhibitor (NRTI) resistance
* Treated with only one previous ART regimen. Single drug substitutions for toxicity, simplification, changes in national guidelines or drug availability are allowed
* At least one NRTI with predicted preserved activity available for a background regimen
* In settings where resistance tests are routinely available, at least one new active NRTI from tenofovir disoproxil fumarate, abacavir or zidovudine should have preserved activity based on cumulative results of resistance tests
* In settings where resistance tests are not routinely available, children who are due to switch according to national guidelines should have at least one new NRTI predicted to be available from tenofovir disoproxil fumarate, abacavir or zidovudine
* Viral load ≥ 500 c/ml at screening visit

Exclusion Criteria:

* History or presence of known allergy or contraindications to dolutegravir
* History or presence of known allergy or contraindications to proposed available NRTI backbone or proposed available SOC third agent.
* Alanine aminotransferase (ALT) ≥ 5 times the upper limit of normal, OR ALT ≥3x upper limit of normal and bilirubin ≥2x upper limit of normal
* Patients with severe hepatic impairment or unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Anticipated need for Hepatitis C virus (HCV) therapy during the study
* Pregnancy or breastfeeding
* Evidence of lack of susceptibility to integrase inhibitors or more than a 2-week exposure to antiretrovirals of this class

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 792 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Gibb, Principal Investigator — Medical Research Council Clinical Trials Unit at UCL
Locations (28):
- Germany (2):
  - Universitata Frankfurt, Frankfurt
  - UkE Eppendorf Hamburg, Hamburg
- Centro Materno-Infantil de Norte, Porto, Portugal
- South Africa (5):
  - King Edward VIII Hospital, Durban
  - Africa Health Research Institute (AHRI), Hlabisa
  - PHRU Klerksdorp, Klerksdorp
  - Kid-Cru, Parow
  - PHRU, Soweto
- Spain (3):
  - Hospital San Joan de Defu, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
- Thailand (6):
  - Prapokklao Hospital, Chanthaburi
  - Nakornping Hospital, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Khon Kaen Hospital, Khon Kaen
  - Mahasarakam Hospital, Maha Sarakham
  - Phayao Hospital, Phayao
- Uganda (4):
  - Baylor, Kampala
  - JCRC, Kampala
  - MUJHU, Kampala
  - JCRC, Mbarara
- United Kingdom (6):
  - Birmingham Heartlands Hospital, Birmingham
  - Leeds General Infirmary, Leeds
  - Leicester Royal Infirmary, Leicester
  - Great Ormand Street Hospital, London
  - Kings College Hospital, London
  - St Mary's Hospital, London
- UZCRC, Harare, Zimbabwe

REFERENCES:
- [Result] Turkova A, White E, Mujuru HA, Kekitiinwa AR, Kityo CM, Violari A, Lugemwa A, Cressey TR, Musoke P, Variava E, Cotton MF, Archary M, Puthanakit T, Behuhuma O, Kobbe R, Welch SB, Bwakura-Dangarembizi M, Amuge P, Kaudha E, Barlow-Mosha L, Makumbi S, Ramsagar N, Ngampiyaskul C, Musoro G, Atwine L, Liberty A, Musiime V, Bbuye D, Ahimbisibwe GM, Chalermpantmetagul S, Ali S, Sarfati T, Wynne B, Shakeshaft C, Colbers A, Klein N, Bernays S, Saidi Y, Coelho A, Grossele T, Compagnucci A, Giaquinto C, Rojo P, Ford D, Gibb DM; ODYSSEY Trial Team. Dolutegravir as First- or Second-Line Treatment for HIV-1 Infection in Children. N Engl J Med. 2021 Dec 30;385(27):2531-2543. doi: 10.1056/NEJMoa2108793. PMID 34965338
- [Result] Amuge P, Lugemwa A, Wynne B, Mujuru HA, Violari A, Kityo CM, Archary M, Variava E, White E, Turner RM, Shakeshaft C, Ali S, Nathoo KJ, Atwine L, Liberty A, Bbuye D, Kaudha E, Mngqibisa R, Mosala M, Mumbiro V, Nanduudu A, Ankunda R, Maseko L, Kekitiinwa AR, Giaquinto C, Rojo P, Gibb DM, Turkova A, Ford D; ODYSSEY Trial Team. Once-daily dolutegravir-based antiretroviral therapy in infants and children living with HIV from age 4 weeks: results from the below 14 kg cohort in the randomised ODYSSEY trial. Lancet HIV. 2022 Sep;9(9):e638-e648. doi: 10.1016/S2352-3018(22)00163-1. PMID 36055295
- [Derived] Turkova A, White E, Violari A, Mujuru HA, Kekitiinwa AR, Lugemwa A, Kaudha E, Na-Rajsima S, Ahimbisibwe GM, Variavae E, Archary M, Akhalwaya Y, Puthanakit T, Bwakura-Dangarembizi M, Bbuye D, Kasozi M, Liberty A, Konigs C, Welch SB, Riault Y, Bamford A, Cressey TR, Musoke P, Kityo C, Ferrand R, Giaquinto C, Rojo P, Gibb DM, Ford D; ODYSSEY trial team. Weight gain, body composition, and metabolic parameters of dolutegravir-based antiretroviral therapy versus standard of care in children and adolescents: an ancillary analysis of the ODYSSEY trial. Lancet Child Adolesc Health. 2026 Jan 21:S2352-4642(25)00339-6. doi: 10.1016/S2352-4642(25)00339-6. Online ahead of print. PMID 41579881
- [Derived] White E, Kityo C, Spyer MJ, Mujuru HA, Nankya I, Kekitiinwa AR, Lugemwa A, Kaudha E, Liberty A, Cassim H, Archary M, Cotton MF, Ahimbisibwe GM, Cressey TR, Ngampiyaskul C, Srirompotong U, Behuhuma O, Saidi Y, Bamford A, Kobbe R, Nastouli E, Rojo P, Giaquinto C, Gibb DM, Ford D, Turkova A; ODYSSEY trial team. Virological outcomes and genotypic resistance on dolutegravir-based antiretroviral therapy versus standard of care in children and adolescents: a secondary analysis of the ODYSSEY trial. Lancet HIV. 2025 Mar;12(3):e201-e213. doi: 10.1016/S2352-3018(24)00155-3. Epub 2025 Feb 17. PMID 39978387
- [Derived] Barlow-Mosha LN, Ahimbisibwe GM, Chappell E, Amuge PM, Nanduudu A, Kaudha E, Amukele T, Balamusani D, Kafufu B, Nimwesiga A, Kataike H, Namwanje R, Kasangaki G, Mulindwa A, Muzorah GA, Bbuye D, Musiime V, Mujyambere E, Ssenyonga M, Mulima D, Kyambadde RC, Namusanje J, Isabirye R, Nabalamba M, Nakirya BM, Kityo C, Kekitiinwa AR, Giaquinto C, Copp A, Gibb DM, Ford D, Musoke P, Turkova A; ODYSSEY trial team. Effect of dolutegravir on folate, vitamin B12 and mean corpuscular volume levels among children and adolescents with HIV: a sub-study of the ODYSSEY randomized controlled trial. J Int AIDS Soc. 2023 Sep;26(9):e26174. doi: 10.1002/jia2.26174. PMID 37766505
- [Derived] Turkova A, Waalewijn H, Chan MK, Bollen PDJ, Bwakura-Dangarembizi MF, Kekitiinwa AR, Cotton MF, Lugemwa A, Variava E, Ahimbisibwe GM, Srirompotong U, Mumbiro V, Amuge P, Zuidewind P, Ali S, Kityo CM, Archary M, Ferrand RA, Violari A, Gibb DM, Burger DM, Ford D, Colbers A; ODYSSEY Trial Team. Dolutegravir twice-daily dosing in children with HIV-associated tuberculosis: a pharmacokinetic and safety study within the open-label, multicentre, randomised, non-inferiority ODYSSEY trial. Lancet HIV. 2022 Sep;9(9):e627-e637. doi: 10.1016/S2352-3018(22)00160-6. Epub 2022 Jul 19. PMID 35868341
- [Derived] Singh RP, Adkison KK, Baker M, Parasrampuria R, Wolstenholme A, Davies M, Sewell N, Brothers C, Buchanan AM. Development of Dolutegravir Single-entity and Fixed-dose Combination Formulations for Children. Pediatr Infect Dis J. 2022 Mar 1;41(3):230-237. doi: 10.1097/INF.0000000000003366. PMID 34817414
- [Derived] Moore CL, Turkova A, Mujuru H, Kekitiinwa A, Lugemwa A, Kityo CM, Barlow-Mosha LN, Cressey TR, Violari A, Variava E, Cotton MF, Archary M, Compagnucci A, Puthanakit T, Behuhuma O, Saiotadi Y, Hakim J, Amuge P, Atwine L, Musiime V, Burger DM, Shakeshaft C, Giaquinto C, Rojo P, Gibb DM, Ford D; ODYSSEY Trial Team. ODYSSEY clinical trial design: a randomised global study to evaluate the efficacy and safety of dolutegravir-based antiretroviral therapy in HIV-positive children, with nested pharmacokinetic sub-studies to evaluate pragmatic WHO-weight-band based dolutegravir dosing. BMC Infect Dis. 2021 Jan 4;21(1):5. doi: 10.1186/s12879-020-05672-6. PMID 33446115
- [Derived] Bollen PDJ, Moore CL, Mujuru HA, Makumbi S, Kekitiinwa AR, Kaudha E, Parker A, Musoro G, Nanduudu A, Lugemwa A, Amuge P, Hakim JG, Rojo P, Giaquinto C, Colbers A, Gibb DM, Ford D, Turkova A, Burger DM; ODYSSEY trial team. Simplified dolutegravir dosing for children with HIV weighing 20 kg or more: pharmacokinetic and safety substudies of the multicentre, randomised ODYSSEY trial. Lancet HIV. 2020 Aug;7(8):e533-e544. doi: 10.1016/S2352-3018(20)30189-2. PMID 32763217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment to the >=14kg cohort took place between 20th September 2016 and 22nd June 2018 in 8 countries (Germany, Portugal, South Africa, Spain, Thailand, Uganda, United Kingdom, and Zimbabwe) across 29 centres.
  Recruitment to the <14kg cohort took place between 5th July 2018 and 26th August 2019 in the African countries across 7 centres.
  The results published relate to the randomised phase of the study for the >=14kg cohort and <14kg cohort.
Pre-assignment Details: >=14kg: 819 children assessed for eligibility. 109 were ineligible: 102 failed eligibility criteria, 3 didn't return in window and 4 other reasons. Also, 3 children randomised in error: 1 not ART naïve in ODYSSEY A and 3 randomised before DTG available for weight.
  <14kg: 102 children assessed for eligibility. 17 were ineligible: 14 failed eligibility criteria, 1 died before enrolment, 1 carer declined bloods and 1 ineligible due to no protocol approval at site to recruit <14kg cohort.
Groups:
- Dolutegravir (>=14kg Cohort); Dolutegravir (<14kg Cohort): Experimental arm. DTG + 2 nucleoside transcriptase inhibitors. IMP product Dolutegravir (DTG).
- Standard of Care (>=14kg Cohort); Standard of Care (<14kg Cohort): Active comparator arm.
  SOC for ODYSSEY A is defined as a PI or non nucleoside transcriptase inhibitors + 2 or 3 nucleoside transcriptase inhibitor
  SOC for ODYSSEY B is defined as a PI or non nucleoside transcriptase inhibitor+ 2 nucleoside transcriptase inhibitors
Period: Overall Study
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort)
Started | 350 | 357 | 42 | 43
ODYSSEY A | 154 | 157 | 35 | 37
ODYSSEY B | 196 | 200 | 7 | 6
Completed | 350 | 357 | 42 | 43
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Total
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 792
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 12.2 [9.2 to 15.1] | 12.1 [8.8 to 14.7] | 1.3 [0.5 to 2.0] | 1.5 [0.6 to 2.1] | 11.4 [8.0 to 14.6]
Age, Customized [Count of Participants; unit: Participants]
  <6 months | 0 | 0 | 11 | 8 | 19
  6 months-<1 year | 0 | 0 | 5 | 8 | 13
  1-<2 years | 0 | 0 | 22 | 22 | 44
  2-<6 years | 15 | 11 | 4 | 5 | 35
  6-<12 years | 153 | 164 | 0 | 0 | 317
  12-<18 years | 182 | 182 | 0 | 0 | 364
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 171 | 26 | 18 | 389
  Male | 176 | 186 | 16 | 25 | 403
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African | 310 | 313 | 41 | 42 | 706
  Asian | 28 | 32 | 0 | 0 | 60
  White | 5 | 1 | 0 | 0 | 6
  Other | 7 | 11 | 1 | 1 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 61 | 83 | 8 | 12 | 164
  Uganda | 170 | 161 | 22 | 21 | 374
  Europe | 12 | 13 | 0 | 0 | 25
  Zimbabwe | 79 | 67 | 12 | 10 | 168
  Thailand | 28 | 33 | 0 | 0 | 61
ODYSSEY A/B [Count of Participants; unit: Participants]
  ODYSSEY A (starting first-line ART) | 154 | 157 | 35 | 37 | 383
  ODYSSEY B (Switching to second-line ART) | 196 | 200 | 7 | 6 | 409
Weight [Count of Participants; unit: Participants]
  <6kg | 0 | 0 | 11 | 12 | 23
  6-<10kg | 0 | 0 | 20 | 20 | 40
  10-<14kg | 0 | 0 | 11 | 11 | 22
  14-<20kg | 39 | 43 | 0 | 0 | 82
  20-<25kg | 71 | 64 | 0 | 0 | 135
  25-<30kg | 58 | 59 | 0 | 0 | 117
  30-<35kg | 38 | 51 | 0 | 0 | 89
  35-<40kg | 29 | 32 | 0 | 0 | 61
  >=40kg | 115 | 108 | 0 | 0 | 223
Weight-for-age z-score [Count of Participants; unit: Participants] — z-scores (standard scores) are the number of standard deviations the observed data is above or below the population (z-score of 0 represents the population median). Positive z-scores represent the standard deviations above the median and negative z-scores represent the standard deviations below the median. Weight-for-age Z scores indicate: <-3SD severely underweight; <-2SD moderately underweight; -2 to 2SD healthy weight; >2SD overweight.
  Participants
    <-3 | 4 | 4 | 14 | 13 | 35
    -3-<-2 | 20 | 12 | 7 | 6 | 45
    -2-<0 | 78 | 83 | 18 | 21 | 200
    >=0 | 14 | 19 | 3 | 3 | 39
    missing | 234 | 239 | 0 | 0 | 473
BMI-for-age z-score [Count of Participants; unit: Participants] — z-scores (standard scores) are the number of standard deviations the observed data is above or below the population (z-score of 0 represents the population median). Positive z-scores represent the standard deviations above the median and negative z-scores represent the standard deviations below the median. BMI-for-age Z scores indicate: <-3SD severe thinness; <-2SD thinness; -2 to 1SD healthy weight; >1SD overweight; >2SD obese.
  Participants
    <-3 | 22 | 11 | 3 | 6 | 42
    -3-<-2 | 20 | 28 | 6 | 6 | 60
    -2-<0 | 216 | 219 | 20 | 14 | 469
    >=0 | 92 | 99 | 13 | 17 | 221
    missing | 0 | 0 | 0 | 0 | 0
CD4% [Count of Participants; unit: Participants]
  <15% | 121 | 108 | 7 | 11 | 247
  15-<30% | 152 | 147 | 22 | 18 | 339
  >=30% | 77 | 102 | 12 | 11 | 202
  Missing | 0 | 0 | 1 | 3 | 4
Viral Load copies/mL [Count of Participants; unit: Participants]
  <10,000 | 93 | 123 | 4 | 7 | 227
  10,000-<100,000 | 159 | 158 | 13 | 5 | 335
  >=100,000 | 98 | 75 | 25 | 26 | 224
  Missing | 0 | 1 | 0 | 5 | 6
History of WHO Staging [Count of Participants; unit: Participants] — WHO clinic staging categorises people living with HIV into four clinical stages from stage 1 (asymptomatic), stage 2 (mild symptoms), stage 3 (advanced symptoms) and stage 4 (AIDS), with stage 4 being the worst outcome.
  Participants
    Stage 1-2 | 253 | 265 | 31 | 25 | 574
    Stage 3 | 69 | 60 | 6 | 8 | 143
    Stage 4 | 28 | 32 | 5 | 10 | 75
CD4 [Count of Participants; unit: Participants]
  <200 cells/mm^3 | 88 | 70 | 3 | 4 | 165
  200 to <500 cells/mm^3 | 118 | 114 | 2 | 3 | 237
  >=500 cells/mm^3 | 144 | 173 | 36 | 33 | 386
  Missing | 0 | 0 | 1 | 3 | 4
Weight [Median (Inter-Quartile Range); unit: kilogram(s)] | 30.4 [23.7 to 43.7] | 31.0 [23.3 to 42.7] | 8.1 [5.6 to 10.0] | 8.2 [5.2 to 10.3] | 28.7 [20.9 to 41.5]
Weight-for-age z-score [Median (Inter-Quartile Range); unit: z-score] — z-scores (standard scores) are the number of standard deviations the observed data is above or below the population (z-score of 0 represents the population median). Positive z-scores represent the standard deviations above the median and negative z-scores represent the standard deviations below the median. Weight-for-age Z scores indicate: <-3SD severely underweight; <-2SD moderately underweight; -2 to 2SD healthy weight; >2SD overweight. Population: Row population differs differs from overall given that weight-for-age Z scores only estimated for participants aged 10 and below.
  z-score
    number analyzed (Participants) | 116 | 118 | 42 | 43 | 319
    (all) | -1.2 [-1.9 to -0.2] | -0.9 [-1.6 to -0.2] | -2.1 [-3.4 to -1.3] | -1.8 [-3.7 to -0.8] | -1.2 [-2.0 to -0.4]
BMI-for-age z-score [Median (Inter-Quartile Range); unit: z-score] — z-scores (standard scores) are the number of standard deviations the observed data is above or below the population (z-score of 0 represents the population median). Positive z-scores represent the standard deviations above the median and negative z-scores represent the standard deviations below the median. BMI-for-age Z scores indicate: <-3SD severe thinness; <-2SD thinness; -2 to 1SD healthy weight; >1SD overweight; >2SD obese.
  z-score | -0.6 [-1.4 to 0.0] | -0.6 [-1.4 to 0.1] | -1.1 [-1.9 to 0.2] | -0.7 [-2.2 to 0.3] | -0.6 [-1.4 to 0.1]
CD4% [Median (Inter-Quartile Range); unit: %] — Population: Data on CD4% at baseline were missing for four participants.
  %
    number analyzed (Participants) | 350 | 357 | 41 | 40 | 788
    (all) | 20 [11 to 29] | 22 [13 to 31] | 24 [17 to 35] | 23 [14 to 30] | 21 [12 to 30]
CD4 [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Data on CD4 at baseline were missing for four participants.
  cells/mm^3
    number analyzed (Participants) | 350 | 357 | 41 | 40 | 788
    (all) | 444 [196 to 652] | 486 [254 to 751] | 1639 [1026 to 2327] | 1221 [633 to 1870] | 494 [248 to 814]
Log 10 Viral load copies/mL [Median (Inter-Quartile Range); unit: copies/mL] — Population: Data on viral load at baseline were missing for six participants.
  copies/mL
    number analyzed (Participants) | 350 | 356 | 42 | 38 | 786
    (all) | 4.5 [3.9 to 5.1] | 4.4 [3.7 to 4.9] | 5.2 [4.4 to 5.8] | 5.4 [4.8 to 5.9] | 4.5 [3.9 to 5.1]

OUTCOME MEASURES:

1. Primary Outcome: Difference in Proportion With Failure (Clinical or Virological)
Description: Treatment failure by 96 weeks.
  Estimated using time to the first occurrence of any of the following components:
  * Insufficient virological response defined as < 1 log10 drop at week 24 and switch to second/third line ART for treatment failure
  * Viral Load (VL)>400 c/ml at or after 36 weeks confirmed by next visit
  * Death due to any cause
  * Any new or recurrent AIDS defining event (WHO 4) or severe WHO 3 events, adjudicated by the Endpoint Review Committee
Time Frame: 96 weeks post randomisation
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Count of Participants; unit: Participants
Groups:
- Dolutegravir - ODYSSEY A (>=14kg Cohort): Experimental arm. DTG + 2 nucleoside transcriptase inhibitors. IMP product Dolutegravir (DTG). ODYSSEY A: Children starting first-line ART
- Standard of Care - ODYSSEY A (>=14kg Cohort): Active comparator arm. ODYSSEY A: children starting first-line ART
  SOC for ODYSSEY A is defined as a PI or non nucleoside transcriptase inhibitors + 2 or 3 nucleoside transcriptase inhibitor
- Dolutegravir - ODYSSEY B (>=14kg Cohort): Experimental arm. DTG + 2 nucleoside transcriptase inhibitors. IMP product Dolutegravir (DTG). ODYSSEY B: children starting second-line ART.
- Standard of Care - ODYSSEY B (>=14kg Cohort): Active comparator arm. ODYSSEY B: children starting second-line ART.
  SOC for ODYSSEY B is defined as a PI or non nucleoside transcriptase inhibitor+ 2 nucleoside transcriptase inhibitors
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 154 | 157 | 196 | 200
Participants
  Insufficient virological response | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 1
  Confirmed VL>=400 copies/mL | 40 | 64 | 9 | 16 | 10 | 26 | 30 | 38
  Severe WHO 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  WHO 4 | 7 | 5 | 1 | 1 | 5 | 5 | 2 | 0
  Death | 0 | 2 | 2 | 4 | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Primary: Diff in adj. KM estimates (>=14kg) Number of subjects included in analysis: 707 Analysis specification: Pre-specified; Test type: Non-Inferiority — >=14kg cohort: Non-inferiority margin 10% in total population and 12% in ODYSSEY A/ODYSSEY B. <14kg cohort: power for efficacy was not prespecified for this cohort; p = 0.004, Bootstrap method; Risk Difference (RD) = -0.08, 95% CI 2-sided [-0.14 to -0.03] — The probability of having virological or clinical treatment failure by 96 weeks (primary endpoint) was estimated using Kaplan-Meier curves adjusted for stratification factors
Statistical Analysis 2: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Statistical Analysis Title: Diff in adj. KM estimates (Frequentist <14kg) Number of subjects included in analysis: 85 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.057, Bootstrap method; Risk Difference (RD) = -0.18, 95% CI 2-sided [-0.36 to 0.02] — The probability of having virological or clinical treatment failure by 96 weeks (primary endpoint) was estimated using Kaplan-Meier curves adjusted for trial cohort (ODYSSEY A or ODYSSEY B)
Statistical Analysis 3: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Statistical Analysis Title: Primary: diff in adj. KM estimates (Bayesian <14kg) Number of subjects included in analysis: 85 Analysis Specification: Pre-specified; Test type: Non-Inferiority — Bayesian estimation was used for the primary analysis of the difference in treatment failure by 96 weeks by arm in <14kg cohort. An informative prior distribution was used based on the treatment effect observed in >=14kg cohort, with relative weight defined by clinical opinion, solicited prior to the main trial results; p = 0.02, Bootstrap method; Risk Difference (RD) = -0.1, 95% CI 2-sided [-0.19 to -0.02] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); Statistical Analysis Title: Diff in adj. KM estimates (ODYSSEY A>=14kg) Number of subjects included in analysis: 311 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.003, Bootstrap method; Risk Difference (RD) = -0.12, 95% CI 2-sided [-0.21 to -0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Diff in adj. KM estimates (ODYSSEY B >=14kg) Number of subjects included in analysis: 396 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.22, Bootstrap method; Risk Difference (RD) = -0.05, 95% CI 2-sided [-0.12 to 0.03] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: HIV-1 RNA <50c/ml at 96 Weeks
Description: Proportion of children with viral load suppression <50 c/ml at 96 weeks.
Time Frame: 96 weeks post randomisation
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 335 | 330 | 35 | 36 | 146 | 140 | 189 | 192
Participants | 270 | 252 | 27 | 19 | 117 | 113 | 153 | 139
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (>=14kg) Number of subjects included in analysis: 665 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.1377, Regression, Logistic; Risk Difference (RD) = 5, 95% CI 2-sided [-1 to 11]
Statistical Analysis 2: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); Statistical Analysis Title: Adjusted difference (ODYSSEY A >=14kg) Number of subjects included in analysis: 286 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.8895, Regression, Logistic; Risk Difference (RD) = -1, 95% CI 2-sided [-10 to 8]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY B >=14kg) Number of subjects included in analysis: 381 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.0435, Regression, Logistic; Risk Difference (RD) = 9, 95% CI 2-sided [0.4 to 17]
Statistical Analysis 4: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Test type: Superiority; p = 0.021, Regression, Logistic; Risk Difference (RD) = 26, 95% CI 2-sided [6 to 47]

3. Secondary Outcome: HIV-1 RNA <400c/mL at 96 Weeks
Description: Proportion of children with viral load suppression <400 c/ml at 96 weeks
Time Frame: 96 weeks post randomisation
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 337 | 333 | 36 | 36 | 146 | 140 | 191 | 193
Participants | 299 | 285 | 33 | 26 | 129 | 124 | 170 | 161
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (>=14kg) Number of subjects included in analysis: 670 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.2256, Regression, Logistic; Risk Difference (RD) = 3, 95% CI 2-sided [-2 to 8]
Statistical Analysis 2: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.9536, Regression, Logistic; Risk Difference (RD) = 0, 95% CI 2-sided [-8 to 7]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY B >=14kg) Number of subjects included in analysis: 384 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.1104, Regression, Logistic; Risk Difference (RD) = 6, 95% CI 2-sided [-1 to 12]
Statistical Analysis 4: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Test type: Superiority; p = 0.038, Regression, Logistic; Risk Difference (RD) = 19, 95% CI 2-sided [2 to 37]

4. Secondary Outcome: Mean Change in CD4 Count From Baseline to Week 96
Description: Reporting mean change from the global baseline value across both arms.
Time Frame: 96 weeks post randomisation
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Mean (Standard Error); unit: cells/mm^3
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 154 | 157 | 196 | 200
cells/mm^3 | 265 (17) | 230 (17) | 72 (116) | 51 (118) | 311 (23) | 267 (24) | 228 (24) | 202 (24)
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (>=14kg) Statistical analysis description: Linear regression of CD4 at week 96, adjusted for randomised arm, baseline CD4 and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 707 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.144, Regression, Linear; Mean Difference (Final Values) = 35, 95% CI 2-sided [-12 to 82]
Statistical Analysis 2: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY A >=14kg) Statistical analysis description: Linear regression of CD4 at week 96, adjusting for randomised arm, baseline CD4 and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 311 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.185, Regression, Linear; Mean Difference (Final Values) = 44, 95% CI 2-sided [-21 to 109]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY B >=14kg) Statistical analysis description: Linear regression of CD4 at week 96, adjusting for randomised arm, baseline CD4 and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 396 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.427, Regression, Linear; Mean Difference (Final Values) = 27, 95% CI 2-sided [-39 to 93]
Statistical Analysis 4: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Test type: Superiority; p = 0.86, Regression, Linear; Median Difference (Final Values) = 30, 95% CI 2-sided [-308 to 368]

5. Secondary Outcome: Mean Change in Total Cholesterol From Baseline to Week 96
Description: Reporting mean change from global baseline value across both arms.
Time Frame: 96 weeks post randomisation
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 154 | 157 | 196 | 200
mg/dl | -5.0 (1.5) | 9.9 (1.5) | 4.5 (5.6) | 29.6 (5.9) | 2.1 (2.3) | 19.6 (2.3) | -10.5 (1.8) | 2.8 (1.8)
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (>=14kg) Statistical analysis description: Linear regression of total cholesterol at week 96, adjusting for randomised arm, baseline total cholesterol and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 707 Analysis Specification: Pre-specified; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Final Values) = -15.1, 95% CI 2-sided [-19 to -11.1]
Statistical Analysis 2: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Statistical Analysis Title: Adjusted Difference (<14kg) Statistical analysis description: Linear regression of total cholesterol at week 96, adjusting for randomised arm, baseline total cholesterol and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 85 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.0032, Regression, Linear; Mean Difference (Final Values) = -24.4, 95% CI 2-sided [-40.3 to -8.5]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY A >=14kg) Statistical analysis description: Linear regression of total cholesterol at week 96, adjusting for randomised arm, baseline total cholesterol and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 311 Analysis Specification: Pre-specified; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Final Values) = -17.5, 95% CI 2-sided [-23.9 to -11.1]
Statistical Analysis 4: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY B >=14kg) Statistical analysis description: Linear regression of total cholesterol at week 96, adjusting for randomised arm, baseline total cholesterol and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 396 Analysis Specification: Pre-specified; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Final Values) = -13.4, 95% CI 2-sided [-18.5 to -8.4]

6. Secondary Outcome: Serious Adverse Events
Description: Incidence of serious adverse events
Time Frame: Randomised phase: follow-up was censored when the last participant reached 96 weeks of follow-up (142 weeks (IQR:124 to 159) in ≥14kg cohort and 124 weeks (112 to 137) in <14kg cohort).
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Number; unit: participants with events
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 154 | 157 | 196 | 200
participants with events | 35 | 40 | 11 | 11 | 23 | 27 | 12 | 13
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Adjusted time to first event (>=14kg) Number of subjects included in analysis: 707 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.53, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.55 to 1.36]
Statistical Analysis 2: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Statistical Analysis Title: Adjusted time to first event (<14kg) Number of subjects included in analysis: 85 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.86, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.47 to 2.49]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); Statistical Analysis Title: Adjusted time to first event (ODYSSEY A >=14kg) Number of subjects included in analysis: 311 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.52, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.48 to 1.46]
Statistical Analysis 4: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Adjusted time to first event (ODYSSEY B >=14kg) Number of subjects included in analysis: 396 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.86, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.42 to 2.04]

7. Secondary Outcome: Grade 3 or Above Clinical and Laboratory Adverse Events
Description: Incidence of new clinical and laboratory grade 3 and 4 adverse events
Time Frame: as for outcome 6
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Number; unit: participants with events
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 154 | 157 | 196 | 200
participants with events | 73 | 86 | 19 | 21 | 48 | 43 | 25 | 43
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.24, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.61 to 1.13]
Statistical Analysis 2: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = 0.83, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.5 to 1.74]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p = 0.57, Regression, Cox; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.75 to 1.7]
Statistical Analysis 4: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.33 to 0.88]

8. Secondary Outcome: Adverse Events Leading to ART Modification Any Grade
Description: Incidence of adverse events (of any grade) leading to treatment modification
Time Frame: Randomised Phase
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Number; unit: participants with events
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 154 | 157 | 196 | 200
participants with events | 5 | 17 | 0 | 2 | 3 | 8 | 2 | 9
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.11 to 0.77]
Statistical Analysis 2: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p = 0.13, Regression, Cox; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.09 to 1.33]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p = 0.055, Regression, Cox; Hazard Ratio (HR) = 0.22, 95% CI 2-sided [0.05 to 1.03]

9. Secondary Outcome: Treatment Failure by 48 Weeks
Description: Treatment failure by 48 weeks. Difference in proportion with clinical or virological failure (as defined above)
Time Frame: 48 weeks post randomisation
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 154 | 157 | 196 | 200
Participants
  Insufficient virologic response | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 1
  Confirmed viral load >400c/ml | 13 | 31 | 4 | 11 | 4 | 12 | 9 | 19
  Severe WHO stage 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  WHO stage 4 | 7 | 5 | 1 | 1 | 5 | 5 | 2 | 0
  Death | 0 | 2 | 2 | 3 | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Diff in adj. KM estimates (>=14kg) Statistical analysis description: Difference in adjusted (for stratification factors) Kaplan-Meier survival function estimates at 48 weeks after randomisation. Number of subjects included in analysis: 707 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.003, Bootstrap method; Risk Difference (RD) = -0.06, 95% CI 2-sided [-0.1 to -0.02] — The probability of having virological or clinical treatment failure by 48 weeks was estimated using Kaplan-Meier curves adjusted for stratification factors
Statistical Analysis 2: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); Statistical Analysis Title: Diff in adj. KM estimates (ODYSSEY A >=14kg) Statistical analysis description: Difference in adjusted (for stratification factors) Kaplan-Meier survival function estimates at 48 weeks after randomisation. Number of subjects included in analysis: 311 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.035, Bootstrap method; Risk Difference (RD) = -0.07, 95% CI 2-sided [-0.13 to -0.01] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Diff in adj. KM estimates (ODYSSEY B >=14kg) Statistical analysis description: Difference in adjusted (for stratification factors) Kaplan-Meier survival function estimates at 48 weeks after randomisation. Number of subjects included in analysis: 396 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.039, Bootstrap method; Risk Difference (RD) = -0.05, 95% CI 2-sided [-0.11 to -0.004] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.057, Other [Bootstrap method]; Risk Difference (RD) = -0.18, 95% CI 2-sided [-0.36 to 0.02]

10. Secondary Outcome: Treatment Failure by 144 Weeks
Description: Treatment failure by 144 weeks. Difference in proportion with clinical or virological failure (as defined above)
Time Frame: 144 weeks post randomisation
Population: Note: analysis could not be performed in <14kg cohort due to shorter follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 154 | 157 | 196 | 200
Participants
  Insufficient virologic response | 0 | 3 | 0 | 2 | 0 | 1
  Confirmed viral load>400c/mL | 48 | 76 | 13 | 28 | 35 | 48
  Severe WHO stage 3 | 0 | 1 | 0 | 0 | 0 | 1
  WHO stage 4 | 8 | 5 | 6 | 5 | 2 | 0
  Death | 0 | 2 | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Diff in adj. KM estimates (>=14kg) Statistical analysis description: Difference in adjusted (for stratification factors) Kaplan-Meier survival function estimates at 144 weeks after randomisation. Number of subjects included in analysis: 707 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.003, Bootstrap method; Risk Difference (RD) = -0.09, 95% CI 2-sided [-0.16 to -0.04] — The probability of having virological or clinical treatment failure by 144 weeks was estimated using Kaplan-Meier curves adjusted for stratification factors
Statistical Analysis 2: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); Statistical Analysis Title: Diff in adj. KM estimates (ODYSSEY A >=14kg) Statistical analysis description: Difference in adjusted (for stratification factors) Kaplan-Meier survival function estimates at 144 weeks after randomisation. Number of subjects included in analysis: 311 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.009, Bootstrap method; Risk Difference (RD) = -0.12, 95% CI 2-sided [-0.21 to -0.03] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Diff in adj. KM estimates (ODYSSEY B >=14kg) Statistical analysis description: Difference in adjusted (for stratification factors) Kaplan-Meier survival function estimates at 144 weeks after randomisation. Number of subjects included in analysis: 396 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.079, Bootstrap method; Risk Difference (RD) = -0.08, 95% CI 2-sided [-0.16 to 0.01] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: WHO 4, Severe WHO 3 Events and Death
Description: Rate of clinical events : WHO 4, severe WHO 3 events and death
Time Frame: as for outcome 6
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 154 | 157 | 196 | 200
Participants | 8 | 8 | 3 | 6 | 6 | 6 | 2 | 2
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.993, Regression, Cox; Hazard Ratio (HR) = 1, 95% CI 2-sided [0.38 to 2.68]
Statistical Analysis 2: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = 0.33, Regression, Cox; Hazard Ratio (HR) = 0.5, 95% CI 2-sided [0.13 to 2]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p = 0.991, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.32 to 3.12]
Statistical Analysis 4: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p = 0.997, Regression, Cox; Hazard Ratio (HR) = 1, 95% CI 2-sided [0.14 to 7.13]

12. Secondary Outcome: Per Protocol: Treatment Failure by 96 Weeks
Description: Per protocol: treatment failure by 96 weeks post randomisation
Time Frame: 96 weeks post randomisation
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 340 | 337 | 42 | 43 | 150 | 145 | 190 | 192
Participants | 44 | 62 | 12 | 20 | 13 | 28 | 31 | 34
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Diff in adj. KM estimates (>=14kg) Statistical analysis description: Difference in adjusted (for stratification factors) Kaplan-Meier survival function estimates at 96 weeks after randomisation. Number of subjects included in analysis: 677 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.015, Bootstrap method; Risk Difference (RD) = -0.07, 95% CI 2-sided [-0.12 to -0.01] — The probability of having virological or clinical treatment failure by 96 weeks (per protocol analysis) was estimated using Kaplan-Meier curves adjusted for stratification factors
Statistical Analysis 2: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Statistical Analysis Title: Adjusted difference (frequentist <14kg) Statistical analysis description: Difference in adjusted (for stratification factors) Kaplan-Meier survival function estimates at 96 weeks after randomisation. Number of subjects included in analysis: 85 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.075, Bootstrap method; Risk Difference (RD) = -0.172, 95% CI 2-sided [-0.362 to 0.029] — The probability of having virological or clinical treatment failure by 96 weeks (per protocol analysis) was estimated using Kaplan-Meier curves adjusted for trial cohort (ODYSSEY A or ODYSSEY B)
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY A >=14kg) Statistical analysis description: Difference in adjusted (for stratification factors) Kaplan-Meier survival function estimates at 96 weeks after randomisation. Number of subjects included in analysis: 295 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.004, Bootstrap method; Risk Difference (RD) = -0.126, 95% CI 2-sided [-0.21 to -0.036] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY B >=14kg) Statistical analysis description: Difference in adjusted (for stratification factors) Kaplan-Meier survival function estimates at 96 weeks after randomisation. Number of subjects included in analysis: 382 Analysis Specification: Pre-specified; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.547, Bootstrap method; Risk Difference (RD) = -0.023, 95% CI 2-sided [-0.096 to 0.056] — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Any Drug Class Resistance After Virologic Failure
Description: Any drug class resistance after virologic failure 96 weeks post randomisation
  Major International AIDS Society (IAS) drug-resistance mutations were defined according to the 2019 update of the IAS drug-resistance mutations.
Time Frame: 96 weeks post randomisation
Population: Shown are the numbers of participants with resistance after virologic failure, among those with virologic failure by week 96 who had a post-treatment failure resistance test available for the drug class.
Measure: Count of Participants; unit: Participants
Groups:
- Dolutegravir - ODYSSEY A (<14kg Cohort): Experimental arm. DTG + 2 nucleoside transcriptase inhibitors. IMP product Dolutegravir (DTG). ODYSSEY A: Children starting first-line ART
- Standard of Care - ODYSSEY A (<14kg Cohort): Active comparator arm. ODYSSEY A: children starting first-line ART SOC for ODYSSEY A is defined as a PI or non nucleoside transcriptase inhibitors + 2 or 3 nucleoside transcriptase inhibitor
- Dolutegravir - ODYSSEY B (<14kg Cohort): Experimental arm. DTG + 2 nucleoside transcriptase inhibitors. IMP product Dolutegravir (DTG). ODYSSEY B: children starting second-line ART.
- Standard of Care - ODYSSEY B (<14kg Cohort): Active comparator arm. ODYSSEY B: children starting second-line ART. SOC for ODYSSEY B is defined as a PI or non nucleoside transcriptase inhibitor+ 2 nucleoside transcriptase inhibitors
Arm/Group | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort) | Dolutegravir - ODYSSEY A (<14kg Cohort) | Standard of Care - ODYSSEY A (<14kg Cohort) | Dolutegravir - ODYSSEY B (<14kg Cohort) | Standard of Care - ODYSSEY B (<14kg Cohort)
Number analyzed (Participants) | 11 | 29 | 29 | 40 | 6 | 12 | 2 | 3
Participants | 0 | 28 | 23 | 36 | 6 | 12 | 2 | 3

14. Secondary Outcome: NRTI Resistance After Virologic Failure
Description: NRTI resistance after virologic failure 96 weeks post randomisation.
  Major International AIDS Society (IAS) drug-resistance mutations were defined according to the 2019 update of the IAS drug-resistance mutations.
Time Frame: 96 weeks post randomisation
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort) | Dolutegravir - ODYSSEY A (<14kg Cohort) | Standard of Care - ODYSSEY A (<14kg Cohort) | Dolutegravir - ODYSSEY B (<14kg Cohort) | Standard of Care - ODYSSEY B (<14kg Cohort)
Number analyzed (Participants) | 11 | 29 | 29 | 40 | 6 | 12 | 2 | 3
Participants | 0 | 18 | 21 | 31 | 1 | 10 | 1 | 3

15. Secondary Outcome: NNRTI Resistance After Virologic Failure
Description: NNRTI resistance after virologic failure 96 weeks post randomisation.
  Major International AIDS Society (IAS) drug-resistance mutations were defined according to the 2019 update of the IAS drug-resistance mutations.
Time Frame: 96 weeks post randomisation
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care - ODYSSEY A (<14kg Cohort): Active comparator arm. ODYSSEY A: children starting first-line ART SOC for ODYSSEY A is defined as a PI or non nucleoside transcriptase inhibitors + 2 or 3 nucleoside transcriptase inhibitors
Arm/Group | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort) | Dolutegravir - ODYSSEY A (<14kg Cohort) | Standard of Care - ODYSSEY A (<14kg Cohort) | Dolutegravir - ODYSSEY B (<14kg Cohort) | Standard of Care - ODYSSEY B (<14kg Cohort)
Number analyzed (Participants) | 11 | 29 | 29 | 40 | 6 | 12 | 2 | 3
Participants | 0 | 27 | 22 | 36 | 6 | 11 | 2 | 3

16. Secondary Outcome: PI Resistance After Virologic Failure
Description: PI resistance after virologic failure 96 weeks post randomisation.
  Major International AIDS Society (IAS) drug-resistance mutations were defined according to the 2019 update of the IAS drug-resistance mutations.
Time Frame: 96 weeks post randomisation
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort) | Dolutegravir - ODYSSEY A (<14kg Cohort) | Standard of Care - ODYSSEY A (<14kg Cohort) | Dolutegravir - ODYSSEY B (<14kg Cohort) | Standard of Care - ODYSSEY B (<14kg Cohort)
Number analyzed (Participants) | 11 | 29 | 29 | 40 | 6 | 12 | 2 | 3
Participants | 0 | 0 | 2 | 3 | 0 | 2 | 0 | 0

17. Secondary Outcome: INSTI Resistance After Virologic Failure
Description: INSTI resistance after virologic failure 96 weeks post randomisation
  Major International AIDS Society (IAS) drug-resistance mutations were defined according to the 2019 update of the IAS drug-resistance mutations.
Time Frame: 96 weeks post randomisation
Population: Shown are the numbers of participants with resistance after virologic failure, among those with virologic failure by week 96 who had a post-treatment failure resistance test available for the drug class. The integrase gene was not sequenced for standard of care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Dolutegravir - ODYSSEY A (<14kg Cohort) | Dolutegravir - ODYSSEY B (<14kg Cohort)
Number analyzed (Participants) | 11 | 22 | 5 | 2
Participants | 0 | 4 | 0 | 1

18. Secondary Outcome: Emerging Resistance to Any Drug Class After Virologic Failure
Description: Emerging resistance to any drug class after virologic failure 96 weeks post randomisation
  Major International AIDS Society (IAS) drug-resistance mutations were defined according to the 2019 update of the IAS drug-resistance mutations.
  >=14kg cohort: among participants with virologic failure and exposure to the drug class, percentage of participants with emerging resistance was estimated under an assumption of the same proportion of new resistance in participants with an available baseline resistance test and those without.
  <14kg cohort: percentage reported for participants with whom resistance test was available post-failure and at baseline, and exposed to drug-class during trial.
Time Frame: 96 weeks post randomisation
Population: Dolutegravir - ODYSSEY A (>=14kg cohort): 0 participants had resistance to INSTI post failure Standard of Care - ODYSSEY B (<14kg Cohort) - 0 participants with virological failure and any gene sequenced at baseline and post-failure.
Measure: Number; unit: percentage of participants
Arm/Group | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort) | Dolutegravir - ODYSSEY A (<14kg Cohort) | Standard of Care - ODYSSEY A (<14kg Cohort) | Dolutegravir - ODYSSEY B (<14kg Cohort) | Standard of Care - ODYSSEY B (<14kg Cohort)
Number analyzed (Participants) | 0 | 21 | 6 | 6 | 5 | 5 | 2 | 0
percentage of participants |  | 97 | 22 | 19 | 0 | 100 | 50 |

19. Secondary Outcome: NRTI Emerging Resistance After Virologic Failure
Description: NRTI emerging resistance after virologic failure 96 weeks post randomisation
  Major International AIDS Society (IAS) drug-resistance mutations were defined according to the 2019 update of the IAS drug-resistance mutations.
  >=14kg cohort: among participants with virologic failure and exposure to the drug class, percentage of participants with emerging resistance was estimated under an assumption of the same proportion of new resistance in participants with an available baseline resistance test and those without.
  <14kg cohort: percentage reported for participants with whom a resistance test was available post-failure and at baseline, and exposed to drug-class during trial.
Time Frame: 96 weeks post randomisation
Population: Dolutegravir - ODYSSEY A (>=14kg cohort) - 0 participants had resistance post failure.
  Dolutegravir - ODYSSEY A (<14kg Cohort) and Standard of Care - ODYSSEY B (<14kg Cohort) - 0 participants with virological failure, exposed to drug-class, and gene sequenced at baseline and post-failure.
Measure: Number; unit: percentage of participants
Arm/Group | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort) | Dolutegravir - ODYSSEY A (<14kg Cohort) | Standard of Care - ODYSSEY A (<14kg Cohort) | Dolutegravir - ODYSSEY B (<14kg Cohort) | Standard of Care - ODYSSEY B (<14kg Cohort)
Number analyzed (Participants) | 0 | 13 | 2 | 3 | 0 | 5 | 1 | 0
percentage of participants |  | 62 | 8 | 10 |  | 100 | 100 |

20. Secondary Outcome: NNRTI Emerging Resistance After Virologic Failure
Description: NNRTI emerging resistance after virologic failure 96 weeks post randomisation
  Major International AIDS Society (IAS) drug-resistance mutations were defined according to the 2019 update of the IAS drug-resistance mutations.
  >=14kg cohort: among participants with virologic failure and exposure to the drug class, percentage of participants with emerging resistance was estimated under an assumption of the same proportion of new resistance in participants with an available baseline resistance test and those without.
  <14kg cohort: percentage reported for participants with whom a resistance test was available post-failure and at baseline, and exposed to drug-class during trial.
Time Frame: 96 weeks post randomisation
Population: Emergent drug resistance estimated only in participants exposed to drug class during trial (DTG arm not exposed to NNRTI class).
  Standard of Care - ODYSSEY A (<14kg Cohort) and Standard of Care - ODYSSEY B (<14kg Cohort) - 0 participants with virological failure, exposed to drug-class, and gene sequenced at baseline and post-failure.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY A (<14kg Cohort) | Standard of Care - ODYSSEY B (<14kg Cohort)
Number analyzed (Participants) | 19 | 2 | 0 | 0
percentage of participants | 88 | 100 |  |

21. Secondary Outcome: PI Emerging Resistance After Virologic Failure
Description: PI emerging resistance after virologic failure 96 weeks post randomisation
  Major International AIDS Society (IAS) drug-resistance mutations were defined according to the 2019 update of the IAS drug-resistance mutations.
  >=14kg cohort: among participants with virologic failure and exposure to the drug class, percentage of participants with emerging resistance was estimated under an assumption of the same proportion of new resistance in participants with an available baseline resistance test and those without.
  <14kg cohort: percentage reported for participants with whom a resistance test was available post-failure and at baseline, and exposed to drug-class during trial.
Time Frame: 96 weeks post randomisation
Population: Emergent drug resistance estimated only in participants exposed to drug class during trial (DTG arm not exposed to PI class).
  Standard of Care - ODYSSEY A (>=14kg cohort) - 0 participants had resistance post failure.
  Standard of Care - ODYSSEY B (<14kg Cohort) - 0 participants with virological failure, exposed to drug-class, and gene sequenced at baseline and post-failure.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY A (<14kg Cohort) | Standard of Care - ODYSSEY B (<14kg Cohort)
Number analyzed (Participants) | 0 | 2 | 1 | 0
percentage of participants |  | 5 | 100 |

22. Secondary Outcome: INSTI Emerging Resistance After Virologic Failure
Description: INSTI emerging resistance after virologic failure 96 weeks post randomisation
  Major International AIDS Society (IAS) drug-resistance mutations were defined according to the 2019 update of the IAS drug-resistance mutations.
  >=14kg cohort: among participants with virologic failure and exposure to the drug class, percentage of participants with emerging resistance was estimated under an assumption of the same proportion of new resistance in participants with an available baseline resistance test and those without.
  <14kg cohort: percentage reported for participants with whom a resistance test was available post-failure and at baseline, and exposed to drug-class during trial.
  The integrase gene was not sequenced for the standard of care arm.
Time Frame: 96 weeks post randomisation
Population: Emergent drug resistance estimated only in participants exposed to drug class during trial (SOC arm not exposed to INSTI drug class).
  Dolutegravir - ODYSSEY A (>=14kg cohort) - 0 participants had resistance post failure.
Measure: Number; unit: percentage of participants
Arm/Group | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Dolutegravir - ODYSSEY A (<14kg Cohort) | Dolutegravir - ODYSSEY B (<14kg Cohort)
Number analyzed (Participants) | 0 | 4 | 5 | 2
percentage of participants |  | 18 | 0 | 50

23. Secondary Outcome: Time to Any New or Recurrent AIDS Defining Event (WHO 4) or Severe WHO 3 Events
Description: Time to any new or recurrent AIDS defining event (WHO 4) or severe WHO 3 events adjudicated by the Endpoint Review Committee.
  Reported in >=14kg and <14kg papers. >=14kg cohort paper (https://www.nejm.org/doi/full/10.1056/NEJMoa2108793) <14kg cohort paper (https://www.thelancet.com/journals/lanhiv/article/PIIS2352-3018(22)00163-1/fulltext)
Time Frame: as for outcome 6
Reporting Status: Not Posted

24. Secondary Outcome: Adherence Questionnaire
Description: The proportion of adherence questionnaires where the participant/carer reports missing a dose within the last week will be compared between randomised groups.
  Reported in >=14kg and <14kg papers. >=14kg cohort paper (https://www.nejm.org/doi/full/10.1056/NEJMoa2108793) <14kg cohort paper (https://www.thelancet.com/journals/lanhiv/article/PIIS2352-3018(22)00163-1/fulltext)
Time Frame: as for outcome 6
Reporting Status: Not Posted

25. Secondary Outcome: Health-related Quality of Life Questionnaire
Description: Adapted from the Euro Quality of Life Questionnaire (Qol)-5D questionnaire The EQ5D-3L (3-level version of EQ-5D) questionnaire contains five questions about the participants' quality of life: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Each question has three dimensions: no problems, some problems, and extreme problems.
  This analysis reports whether the participant reports any problems (some or extreme). Percentages are of participants completing at least one EQ5D-3L questionnaire during follow-up.
  Reported in >=14kg cohort paper (https://www.nejm.org/doi/full/10.1056/NEJMoa2108793)
Time Frame: as for outcome 6
Reporting Status: Not Posted

26. Secondary Outcome: Acceptability Questionnaire
Description: Number of participants reported to have problems with size, taste or swallowing of the medicines as assessed by Acceptability questionnaire
  Reported in >=14kg and <14kg papers. >=14kg cohort paper (https://www.nejm.org/doi/full/10.1056/NEJMoa2108793) <14kg cohort paper (https://www.thelancet.com/journals/lanhiv/article/PIIS2352-3018(22)00163-1/fulltext)
Time Frame: as for outcome 6
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Mean Change in Weight From Baseline
Description: Mean change in weight from baseline to week 96
Time Frame: 96 weeks post randomisation
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Mean (Standard Error); unit: kg
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 154 | 157 | 196 | 200
kg | 7.1 (0.3) | 6.1 (0.3) | 5.0 (0.2) | 5.1 (0.2) | 7.8 (0.4) | 6.5 (0.4) | 6.7 (0.3) | 5.9 (0.3)
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (>=14kg) Number of subjects included in analysis: 707 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.004, Regression, Linear; Mean Difference (Final Values) = 1, 95% CI 2-sided [0.3 to 1.7]
Statistical Analysis 2: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY A >=14kg) Statistical analysis description: Linear regression of weight at week 96, adjusting for randomised arm, baseline weight and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 311 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.024, Regression, Linear; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [0.2 to 2.5]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Adjusting Difference (ODYSSEY B >=14kg) Statistical analysis description: Linear regression of weight at week 96, adjusting for randomised arm, baseline weight and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 396 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.075, Regression, Linear; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.1 to 1.6]
Statistical Analysis 4: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Test type: Superiority; p = 0.67, Regression, Linear; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.8 to 0.5]

28. Other Pre Specified Outcome: Mean Change in BMI-for-age Z-score From Baseline
Description: Mean change in BMI-for-age from baseline to week 96. Reporting mean change from the global baseline value across both arms.
  z-scores (standard scores) are the number of standard deviations the observed data is above or below the population (z-score of 0 represents the population median). Positive z-scores represent the standard deviations above the median and negative z-scores represent the standard deviations below the median. BMI-for-age Z scores indicate: <-3SD severe thinness; <-2SD thinness; -2 to 1SD healthy weight; >1SD overweight; >2SD obese.
Time Frame: 96 weeks post randomisation
Population: Results not presented by ODYSSEY A and B in <14kg cohort due to due ODYSSEY B having too few participants (n=13).
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
Number analyzed (Participants) | 350 | 357 | 42 | 43 | 154 | 157 | 196 | 200
Z-score | 0.24 (0.04) | 0.11 (0.04) | 1.1 (0.3) | 1.5 (0.3) | 0.36 (0.07) | 0.20 (0.07) | 0.14 (0.05) | 0.04 (0.05)
Statistical Analysis 1: Comparison: Dolutegravir (>=14kg Cohort) vs Standard of Care (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (>=14kg) Statistical analysis description: Linear regression of BMI-for-age at week 96, adjusting for randomised arm, baseline BMI-for-age and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 707 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.036, Regression, Linear; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.01 to 0.25]
Statistical Analysis 2: Comparison: Dolutegravir - ODYSSEY A (>=14kg Cohort) vs Standard of Care - ODYSSEY A (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY A >=14kg) Statistical analysis description: Linear regression of BMI-for-age at week 96, adjusting for randomised arm, baseline BMI-for-age and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 311 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.092, Regression, Linear; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.03 to 0.36]
Statistical Analysis 3: Comparison: Dolutegravir - ODYSSEY B (>=14kg Cohort) vs Standard of Care - ODYSSEY B (>=14kg Cohort); Statistical Analysis Title: Adjusted Difference (ODYSSEY B >=14kg) Statistical analysis description: Linear regression of BMI-for-age at week 96, adjusting for randomised arm, baseline BMI-for-age and stratification factors. Presenting mean difference between arms. Number of subjects included in analysis: 396 Analysis Specification: Pre-specified; Test type: Superiority; p = 0.176, Regression, Linear; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.05 to 0.25]
Statistical Analysis 4: Comparison: Dolutegravir (<14kg Cohort) vs Standard of Care (<14kg Cohort); Test type: Superiority; p = 0.50, Regression, Linear; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.1 to 0.5]

ADVERSE EVENTS:
Time Frame: Randomised phase: follow-up was censored when the last participant reached 96 weeks of follow-up (142 weeks (IQR:124 to 159) in ≥14kg cohort and 124 weeks (112 to 137) in <14kg cohort).
Description: Non-serious Adverse Events (AEs):There was no single diagnosis reported for 5% or more of participants. Details of all AEs are reported in the supplementary materials of the >=14kg cohort paper (including by ODYSSEY A/B) (https://www.nejm.org/doi/full/10.1056/NEJMoa2108793) and the <14kg cohort paper (https://www.thelancet.com/journals/lanhiv/article/PIIS2352-3018(22)00163-1/fulltext)
Arm/Group | Dolutegravir (>=14kg Cohort) | Standard of Care (>=14kg Cohort) | Dolutegravir (<14kg Cohort) | Standard of Care (<14kg Cohort) | Dolutegravir - ODYSSEY A (>=14kg Cohort) | Standard of Care - ODYSSEY A (>=14kg Cohort) | Dolutegravir - ODYSSEY B (>=14kg Cohort) | Standard of Care - ODYSSEY B (>=14kg Cohort)
All-Cause Mortality (participants affected / at risk) | 2/350 | 3/357 | 2/42 | 4/43 | 2/154 | 2/157 | 0/196 | 1/200
Serious Adverse Events (participants affected / at risk) | 35/350 | 40/357 | 11/42 | 11/43 | 23/154 | 27/157 | 12/196 | 13/200
Other Adverse Events (participants affected / at risk) | 0/350 | 0/357 | 0/42 | 0/43 | 0/154 | 0/157 | 0/196 | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dolutegravir (>=14kg Cohort) (N=350) | Standard of Care (>=14kg Cohort) (N=357) | Dolutegravir (<14kg Cohort) (N=42) | Standard of Care (<14kg Cohort) (N=43) | Dolutegravir - ODYSSEY A (>=14kg Cohort) (N=154) | Standard of Care - ODYSSEY A (>=14kg Cohort) (N=157) | Dolutegravir - ODYSSEY B (>=14kg Cohort) (N=196) | Standard of Care - ODYSSEY B (>=14kg Cohort) (N=200)
Vascular disorders (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1
Immune system disorders (Immune system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
General disorders and administration site conditions (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Psychiatric disorders (Psychiatric disorders) | 2 | 2 | 0 | 0 | 2 | 2 | 0 | 0
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0
Investigations (Investigations) | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Cardiac disorders (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3 | 3 | 1 | 1 | 1 | 1 | 2 | 2
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders (Nervous system disorders) | 3 | 4 | 0 | 0 | 2 | 4 | 1 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal and urinary disorders (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Infections and infestations (Infections and infestations) | 25 | 23 | 9 | 9 | 19 | 14 | 6 | 9

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT02259127/Prot_SAP_ICF_000.pdf